CLINICAL TRIAL: NCT00957528
Title: The Effects of Cyclic Testosterone Administration on Muscle Function in Older Individuals
Brief Title: Cycled Testosterone Replacement Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01-302; GCRC 615; R01AG022023 (NIH)
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Hypogonadism
Keywords: Low Normal Testosterone; Male; Aging
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; testosterone enanthate; Sesame Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Weekly placebo treatment for a duration of 5 months.
  Interventions: Drug: Placebo
- Monthly Cycled Testosterone (Experimental): A month of weekly testosterone treatment alternated by a month of weekly placebo treatment for a duration of 5 months.
  Interventions: Drug: Testosterone; Drug: Placebo
- Continuous Testosterone (Experimental): Weekly testosterone treatment for a duration of 5 months
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Weekly im injections of 100 mg testosterone enanthate.
  Other Names: Testosterone Enanthate
  Arms: Continuous Testosterone; Monthly Cycled Testosterone
Drug: Placebo — Weekly IM injections of sesame oil.
  Other Names: Sesame Oil
  Arms: Monthly Cycled Testosterone; Placebo

SUMMARY:
The purpose of this study is to determine whether testosterone (male hormone) therapy is effective if administered in a cyclic fashion (periodic dosing) compared to continuous dosing in men aged 60 to 85 years. Effectiveness will be determined based on improvements in body composition, muscle metabolism, muscle strength, and bone metabolism.

DETAILED DESCRIPTION:
Men and women undergo a progressive reduction in lean muscle mass (sarcopenia) with advancing age regardless of their level of physical activity. A 12-yr longitudinal study in healthy sedentary older men showed a correlation between loss of muscle cross-sectional area and muscle strength of the thigh, quadriceps, and flexor muscles. Once weakened, older individuals are prone to falls that prevent independent living and diminish the quality of life. There is a need to develop therapies to counteract losses in skeletal muscle strength with aging. Studies show that exercise and testosterone administration increase skeletal muscle mass and strength in older men. However, the increase in muscle strength by testosterone in older men has not been consistent in all studies. Androgens increase muscle mass by either increasing muscle protein synthesis or inhibiting muscle protein breakdown. This proposal will investigate the hypothesis that cyclic testosterone administration (monthly on/off cycles) will preferentially increase muscle protein synthesis and result in a consistent and greater improvement in muscle strength than continuous testosterone administration.

ELIGIBILITY:
Inclusion Criteria:

* Availability of transportation (i.e., subjects must be able to provide their own transportation to UTMB).

Exclusion Criteria:

* Medications such as anticoagulants (Coumadin) and glucocorticoids.
* History of angina that occurs with exertion or at rest.
* History of myocardial infarction within the last 12 months.
* Failure to successfully complete an exercise stress test using the Bruce protocol. Subjects that demonstrate ≥ 0.1 mV horizontal or downsloping ST segment depression, a drop in systolic blood pressure of ≥ 10 mm Hg, and/or frequent or repetitive arrhythmias (defined as ≥ 10 PVC/min, or couplets) during the stress test will be excluded.
* LDL cholesterol above 200 mg/dL.
* History of prostatic cancer.
* Elevated prostate specific antigen (PSA) above 4.0 µg/L, or severe benign prostatic hypertrophy (BPH) by history (frequent urination, reduced stream).
* Serum total testosterone concentrations of greater than 500 ng/dL.
* Subjects who engage in high intensity, elite training on a regular basis.
* Major medical illness such as diabetes, chronic obstructive pulmonary disease, or sleep apnea.
* Recent history of smoking tobacco.
* Hematocrit greater than 51%.
* Morbidly obese older men (BMI > 35).
* Hypertension: Blood pressure on three consecutive measurements taken at one week intervals that has a systolic pressure ≥ 140 or a diastolic blood pressure ≥ 90. Subjects will be included if they are on two or less blood pressure medications and have a blood pressure below these criteria.
* History of hepatitis or a 3-fold elevation of liver function tests (Alk phos, ALT, AST).
* Bone related disorders such as osteoporosis or parathyroid disease.
* DEXA scans revealing lumbar spine T-scores of less than -2.5.
* Subjects currently taking anti-bone-resorptive agents such as bisphosphonates, parathyroid hormone, or calcitonin.

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Urban, M.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment began in January, 2006 and was closed on December, 2011. Subjects were enrolled at the University of Texas Medical Branch in the Institute for Translational Sciences Clinical Research Center (ITS-CRC).
Pre-assignment Details: Screening was conducted at the ITS-CRC where the subject was consented and screening was conducted to identify eligible subjects.Screening included blood testing and a stress test to determine fitness for physical function testing. Subjects were excluded due to elevated PSA levels, testosterone levels above entry criteria or occult disease.
Period: Overall Study
Arm/Group | Placebo | Monthly Cycled Testosterone | Continuous Testosterone
Started | 8 | 9 | 9
Completed | 8 | 8 | 8
Not Completed | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Monthly Cycled Testosterone | Continuous Testosterone | Total
Number analyzed (Participants) | 8 | 9 | 9 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 2 | 10
  >=65 years | 3 | 6 | 7 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 65.4 (3.22) | 71.6 (7.78) | 73.3 (7.54) | 70.1 (6.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 9 | 9 | 26
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Changes in Basal Muscle Protein Synthesis and Breakdown as Measured by Stable Isotope Metabolic Studies at Baseline and at Five Months
Description: The fractional synthetic rate (FSR) of mixed muscle is calculated by directly measuring the incorporation of L-[ring-13C6]-phenylalanine into protein (%/hr),, using the precursor-product model: FSR = [(EP2 - EP1)/(EM•t)]•60•100, where EP1 and EP2 are the enrichments of bound L-[ring-13C6]-phenylalanine in the first and second muscle biopsies, t is the time interval (min) between biopsies, and EM is the mean L-[ring-13C6]-phenylalanine enrichment in the muscle intracellular pool.
Time Frame: 5 Months
Population: Subjects who completed the entire treatment protocol
Measure: Mean (Standard Deviation); unit: Percent per hour (%/hr)
Arm/Group | Placebo | Monthly Cycled Testosterone | Continuous Testosterone
Number analyzed (Participants) | 8 | 8 | 8
Percent per hour (%/hr)
  Baseline | 0.05 (0.01) | 0.06 (0.01) | 0.06 (0.01)
  Five Months | 0.066 (0.020) | 0.094 (0.014) | 0.101 (0.043)

2. Primary Outcome: Changes in Muscle Strength as Measured by Maximal Voluntary Contraction Tests (Arm Curl) at Baseline, One Month, Two Months, Three Months, Four Months, and at Five Months
Description: Maximum weight (pounds) lifted using Cybex weight machine in a single effort(1-RM) for upper extremities (biceps and triceps) and lower extremities quadriceps and hamstrings).
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Placebo | Monthly Cycled Testosterone | Continuous Testosterone
Number analyzed (Participants) | 8 | 8 | 8
pounds
  Arm Curl Baseline | 39 (12) | 39 (10) | 32 (9)
  Arm Extension Baseline | 40 (9) | 41 (14) | 38 (9)
  Leg Curl Baseline | 46 (6) | 44 (7) | 40 (9)
  Leg Extension Baseline | 70 (21) | 73 (15) | 66 (16)
  Arm Curl Month 1 | 39 (10) | 41 (10) | 34 (8)
  Arm Curl Month 2 | 38 (9) | 40 (10) | 39 (9)
  Arm Curl Month 3 | 39 (9) | 43 (11) | 37 (13)
  Arm Curl Month 4 | 38 (10) | 43 (13) | 41 (12)
  Arm Curl Month 5 | 40 (11) | 45 (13) | 38 (11)
  Arm Extension Month 1 | 40 (7) | 41 (10) | 37 (4)
  Arm Extension Month 2 | 41 (8) | 42 (9) | 44 (10)
  Arm Extension Month 3 | 42 (8) | 43 (7) | 44 (14)
  Arm Extension Month 4 | 42 (8) | 44 (8) | 44 (12)
  Arm Extension Month 5 | 42 (8) | 45 (8) | 45 (10)
  Leg Curl Month 1 | 48 (7) | 46 (9) | 41 (8)
  Leg Curl Month 2 | 51 (11) | 47 (9) | 48 (11)
  Leg Curl Month 3 | 48 (7) | 43 (20) | 48 (14)
  Leg Curl Month 4 | 48 (7) | 50 (10) | 50 (12)
  Leg Curl Month 5 | 48 (10) | 50 (11) | 51 (12)
  Leg Extension Month 1 | 70 (13) | 73 (10) | 67 (15)
  Leg Extension Month 2 | 69 (14) | 77 (16) | 78 (12)
  Leg Extension Month 3 | 74 (13) | 80 (14) | 76 (21)
  Leg Extensuion Month 4 | 72 (14) | 79 (16) | 82 (14)
  Leg Extension Month 5 | 72 (14) | 85 (19) | 83 (17)

3. Primary Outcome: Changes in Lean Body Mass as Measured by Dual Energy X-ray Absorptiometry (DEXA)
Description: Lean body mass is expressed in grams as calculated by Hologic DEXA.
Time Frame: 5 months
Population: All subjects who successfully completed the five month protocol.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Placebo | Monthly Cycled Testosterone | Continuous Testosterone
Number analyzed (Participants) | 8 | 8 | 8
grams
  Lean Body Mass Baseline | 62344 (10368) | 57101 (6671.5) | 57746 (6485.1)
  Lean Body Mass Month 1 | 62994.7 (10308.8) | 59155.4 (6890.9) | 60469.3 (6555.92)
  Lean Body Mass Month 2 | 62038.7 (10556.5) | 56787.8 (6444.16) | 62680.1 (4034.41)
  Lean Body Mass Month 3 | 62256.5 (9881.65) | 59186 (6267.63) | 61167.3 (7530.43)
  Lean Body Mass Month 4 | 62755.4 (10756.2) | 59838.6 (7010.73) | 61436.6 (6997.17)
  Lean Body Month 5 | 61250.6 (11283.3) | 58846.9 (6995.48) | 60871.4 (6840.45)

4. Secondary Outcome: Changes in Bone Mineral Density as Measured by Dual Energy X-ray Absorptiometry (DEXA)
Description: Bone mineral density measure by measured by dual energy x-ray absorptiometry (DEXA)measured at baseline and a five months
Time Frame: 5 months
Measure: Mean (Standard Error); unit: gm/cm^2
Arm/Group | Placebo | Monthly Cycled Testosterone | Continuous Testosterone
Number analyzed (Participants) | 8 | 8 | 8
gm/cm^2
  Total Baseline | 1.12 (0.04) | 1.07 (0.05) | 1.12 (0.05)
  Total Five Months | 1.08 (0.07) | 1.05 (0.05) | 1.14 (0.03)
  Lumbar Spine Baseline | 1.06 (0.07) | 1.00 (0.05) | 1.16 (0.04)
  Lumbar Spine Five Months | 1.07 (0.07) | 1.00 (0.05) | 1.19 (0.06)
  Pelvis baseline | 1.46 (0.16) | 1.15 (0.04) | 1.27 (0.04)
  Pelvis Five Months | 1.28 (0.14) | 1.14 (0.04) | 1.28 (0.06)
  Forearm Baseline | 0.59 (0.02) | 0.59 (0.02) | 0.61 (0.02)
  Forearm Five Months | 0.61 (0.02) | 0.59 (0.03) | 0.62 (0.03)

5. Secondary Outcome: Changes in Serum Markers of Bone Turnover.
Description: Measures of bone turnover markers in serum samples at baseline and at five months.The bone turnover markers analyzed include:
  Markers associated with bone breakdown NTX (N-telopeptide) TRAP5b (tartrate-resistant acid phosphatase isoform 5b) Markers associated with bone formation Osteocalcin BAP (bone specific alkaline phosphatase) Regulators of bone formation iPTH (intact parathyroid hormone) increases in response to bone loss Calcitonin inhibits bone formation in response to elevated levels of serum calcium
Time Frame: 5 months
Measure: Mean (Standard Error); unit: nM BCE (Bone Collagen Equivalents)
Arm/Group | Placebo | Monthly Cycled Testosterone | Continuous Testosterone
Number analyzed (Participants) | 8 | 8 | 8
nM BCE (Bone Collagen Equivalents)
  NTX Baseline | 12 (1.3) | 14 (1.4) | 15 (1.9)
  NTX Five Months | 13 (1.1) | 11 (0.7) | 11 (1.5)
  TRAP5b Baseline | 2 (0.6) | 2 (0.6) | 2 (0.4)
  TRAP5b Five Months | 2 (0.6) | 2 (0.6) | 1 (0.3)
  Osteocalcin Baseline | 8 (0.2) | 8 (0.6) | 9 (0.7)
  Osteocalcin Five Months | 8 (0.5) | 8 (0.5) | 7 (0.8)
  BAP Baseline | 22 (1.5) | 20 (2.3) | 17 (1.5)
  BAP Five Months | 21 (1.3) | 19 (1.9) | 15 (1.7)
  iPTH Baseline | 40 (.3) | 37 (6) | 53 (10)
  iPTH Five Months | 45 (7) | 28 (3) | 60 (15)
  Calcitonin Baseline | 3 (0.4) | 4 (0.6) | 4 (1.3)
  Calcitonin Five months | 3 (0.4) | 4 (0.5) | 3 (0.3)

6. Secondary Outcome: 9473Changes in Serum Inflammatory Biomarkers and Muscle Inflammatory Cytokines
Description: Serum inflammatory biomarkers (Interleukin B-1, 2,5,6,7,8,10,12 13, Interferon gamma, GM-CSF, and Tumor Necrosis Factor alpha)as measured by immunoassay at baseline and at five months
Time Frame: 5 months
Population: All subjects who completed the protocol.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Monthly Cycled Testosterone | Continuous Testosterone
Number analyzed (Participants) | 8 | 8 | 8
pg/mL
  IL-B1 Baseline | 0.14 (0.1) | 0.475 (0.76767) | 1.44143 (2.04769)
  IL-B1 Five Months | 0.20833 (0.22221) | 3.19 (3.24643) | 2.538 (3.33404)
  IL-2 Baseline | 1.32 (1.18655) | 3.19 (3.24643) | 2.538 (3.33404)
  IL-2 Five Months | 2.84 (1.99008) | 1.45333 (0.94076) | 3.862 (5.90798)
  IL-5 Baseline | 0.6 (0.71529) | 0.79 (0.76783) | 1.41875 (1.92013)
  IL-5 Five Months | 0.705 (1.32898) | 0.32286 (0.30065) | 1.94125 (3.46852)
  IL-6 Baseline | 5.68375 (6.78293) | 4.90857 (6.43277) | 10.4025 (20.5897)
  IL-6 Five months | 5.05 (6.0643) | 6.487 (178.673) | 13.89 (28.8691)
  IL-7 Baseline | 8.78 (10.4076) | 11.9688 (16.2135) | 5.19875 (2.84198)
  IL-7 Five Months | 7.68 (10.898) | 23.1888 (52.3705) | 16.2763 (19.6011)
  IL-8 Baseline | 4.5575 (2.67011) | 6.66375 (4.50933) | 8.45625 (11.836)
  IL-8 Five months | 4.3225 (2.0872) | 4.06286 (1.76795) | 11.8025 (20.6936)
  IL-10 Baseline | 22.6363 (41.8883) | 11.2588 (8.19838) | 109.446 (240.088)
  IL-10 Five Months | 25.4525 (41.4135) | 8.34143 (3.65748) | 135.64 (265.7)
  IL-12 Baseline | 7.075 (12.3805) | 4.242 (4.07052) | 35.3583 (56.0444)
  IL-12 Five Months | 10.902 (17.4143) | 2.66 (3.7993) | 58.4217 (86.8424)
  IL-13 baseline | 37.045 (51.9229) | 23.33 (48.7029) | 60.2125 (102.473)
  IL-13 Five Months | 43.465 (61.0587) | 12.72 (17.2687) | 73.674 (148.613)
  IFN gamma Baseline | 10.115 (15.7219) | 4.58 (7.63943) | 23.425 (28.8768)
  IFN gamma Five Months | 36.05 (68.7309) | 1.758 (1.98486) | 36.822 (69.571)
  GM-CSF Baseline | 1.52429 (2.46286) | 2.4 (2.58639) | 7.94875 (16.6389)
  GM-CSF Five Months | 2.27857 (3.19199) | 1.312 (0.88649) | 14.965 (37.1713)
  TNF alpha Baseline | 9.0175 (4.60793) | 10.0863 (4.51058) | 13.215 (10.1743)
  TNF alpha Five Months | 8.14 (3.95778) | 8.1529 (3.70965) | 15.4138 (13.0438)

ADVERSE EVENTS:
Arm/Group | Placebo | Monthly Cycled Testosterone | Continuous Testosterone
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Monthly Cycled Testosterone (N=8) | Continuous Testosterone (N=8)
Saphenous vein clot (Vascular disorders) | 1 | 0 | 1
vertigo (Nervous system disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No